CLINICAL TRIAL: NCT00905567
Title: Randomized, 2-Way Crossover, Bioequivalence Study of Topiramate 25 mg Tablets Administered as 2 x 25 mg Tablets in Healthy Subjects Under Fed Conditions
Brief Title: Topiramate 25 mg Tablets Under Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Pharmaceuticals USA (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 01178
Record Dates: First submitted 2009-05-18; First posted 2009-05-20 (Estimated); Results first posted 2009-09-23 (Estimated); Last update posted 2009-09-23 (Estimated); Status verified 2009-08

CONDITIONS: Healthy
Keywords: Bioequivalence; Healthy Subjects
MeSH Terms: interventions — Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test First (Experimental): Topiramate 2 x 25 mg Tablet
  Interventions: Drug: Topiramate 2 x 25 mg tablet
- Reference First (Active Comparator): Topamax® Tablet 2 x 25 mg
  Interventions: Drug: Topamax® Tablet 2 x 25 mg

INTERVENTIONS:
Drug: Topiramate 2 x 25 mg tablet
  Arms: Test First
Drug: Topamax® Tablet 2 x 25 mg
  Arms: Reference First

SUMMARY:
The objective of this study was to compare the rate and extent of absorption of topiramate 25 mg tablets (test) versus Topamax® (reference) administered as 2 x 25 mg tablets under fed conditions.

DETAILED DESCRIPTION:
Criteria for Evaluation: FDA Bioequivalence Criteria

Statistical Methods: FDA bioequivalence statistical methods

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be females and/or males, non-smokers, 18 years of age or older
* Subjects should read, sign and date an Informed Consent Form prior to any study procedures.
* Female subjects will be post-menopausal or surgically sterilized.
* Post menopausal status is defined as absence of menses for the past 12 months or bilateral oophorectomy at least 6 months ago or hysterectomy with bilateral oophorectomy at least 6 months ago.
* Sterile status is defined as hysterectomy, bilateral oophorectomy or tubal ligation aat least 6 months ago.

Exclusion Criteria:

* Clinically significant illnesses within 4 weeks of the administration of study medication.
* Clinically significant surgery within 4 weeks prior to the administration of the study medication.
* Any history or presence of significant neurological, hepatic, renal, endocrinal, cardiovascular, pulmonary, hematologic, immunologic, psychiatric or metabolic disease.
* Any clinically significant abnormality found during medical screening.
* Abnormal laboratory tests judged clinically significant.
* Positive urine drug screen at screening.
* Positive alcohol breath test at screening.
* Subjects who use tobacco in any form will not be eligible to participate in this study. Three months abstinence is required.
* Positive testing for hepatitis B, hepatitis C or HIV at screening.
* ECG or vital sign abnormalities (clinically significant).
* Subjects with BMI greater than or equal to 30.0.
* History of significant alcohol abuse within 6 months of the screening visit or any indication of the regular use of more than two units of alcohol per day (1 Unit = 150 mL of wine or 360 mL of beer or 45 mL of alcohol 40%).
* History of drug abuse or use of illegal drugs: use of soft drugs (such as marijuana) within 3 months of the screening visit or hard drugs (such as cocaine, phencyclidine (PCP) and crack) within 1 year of the screening visit.
* Any food allergy, intolerance, restriction or special diet that, in the opinion of the medical subinvestigator, contraindicates the subjects participation in this study.
* History of allergic reactions to topiramate.
* Use of any drugs known to induce or inhibit hepatic drug metabolism, use of an investigational drug or participation in an investigational study within 30 days prior to administration of the study medication.
* Use of prescription medication within 14 days prior to administration of study medication or over-the-counter products within 7 days prior to administration of study medication, except for topical products without systemic absorption.
* Donation of plasma (500 mL) within 7 days or donation or significant loss of whole blood (500 mL) within 56 days prior to administration of the study medication.
* Any reason which, in the opinion of the medical subinvestigator, would prevent the subject from participating in the study.

Additional exclusion criteria for females only:

• Positive urine pregnancy test at screening (performed on all females).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2001-06; Primary Completion 2001-06 (Actual); Study Completion 2001-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benoit Girard, MD, Principal Investigator — Anapharm
Locations (1):
- Anapharm Inc., Sainte-Foy, Quebec, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Topiramate (Test) First: Topiramate 2 x 25 mg Tablet (test)dosed in first period followed by Topamax® 2 x 25 mg Tablet (reference) dosed in second period
- Topamax® (Reference) First: Topamax® Tablet 2 x 25 mg (reference) dosed in first period followed by Topiramate 2 x 25 mg Tablet (test) dosed in second period
Period: Period 1
Arm/Group | Topiramate (Test) First | Topamax® (Reference) First
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0
Period: Washout
Arm/Group | Topiramate (Test) First | Topamax® (Reference) First
Started | 12 | 12
Completed | 12 | 11
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Period 2
Arm/Group | Topiramate (Test) First | Topamax® (Reference) First
Started | 12 | 11
Completed | 12 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Topiramate (Test) First | Topamax® (Reference) First | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 12 | 24
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 10 | 9 | 19
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 12 | 12 | 24
Region of Enrollment [Number; unit: participants]
  Canada | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Cmax - Maximum Observed Concentration
Description: Bioequivalence based on Cmax
Time Frame: Blood samples collected over 96 hour period
Population: Data from all subjects who completed the study was included in statistical analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Topiramate: Topiramate 2 x 25 mg Tablet
- Topamax®: Topamax® Tablet 2 x 25 mg
Arm/Group | Topiramate | Topamax®
Number analyzed (Participants) | 23 | 23
ng/mL | 633.96 (251.55) | 700.79 (310.12)
Statistical Analysis 1: Comparison: Topiramate vs Topamax®; Test type: Non-Inferiority or Equivalence — ANOVA was performed on ln-transformed AUC0-t, AUC0-72h, and Cmax. All analyses were performed according to FDA's guidleines; Ratio of the Least Squares Mean = 93.01 — Bioequivalence is established when Ratio of the Least Squares Mean (test/reference x 100) falls within 80-125

2. Primary Outcome: AUC0-72 - Area Under the Concentration Time Curve From Time Zero to Time 72 Hours (Per Participant)
Description: Bioequivalence based on AUC0-72
Time Frame: Blood samples collected over 96 hour period
Population: Data from all subjects who completed the study was included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Topiramate | Topamax®
Number analyzed (Participants) | 23 | 23
ng*hr/mL | 20792.34 (7701.94) | 21930.92 (9118.60)
Statistical Analysis 1: Comparison: Topiramate vs Topamax®; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the Least Squares Mean = 96.62 — Bioequivalence is established when the Ratio of the Least Squares Mean (test/reference x 100) falls within 80-125

3. Primary Outcome: AUC0-t - Area Under the Concentration-time Curve From Time Zero to Time of Last Non-zero Concentration (Per Participant)
Description: Bioequivalence based on AUC0-t
Time Frame: Blood samples collected over 96 hour period
Population: Data from all subjects who completed the study was used in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Topiramate | Topamax®
Number analyzed (Participants) | 23 | 23
ng*hr/mL | 23634.03 (8515.55) | 24918.64 (9927.37)
Statistical Analysis 1: Comparison: Topiramate vs Topamax®; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the Least Squares Mean = 96.43 — Bioequivalence is established when the Ratio of the Least Squares Mean (test/reference x 100) falls within 80-125

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI is not permitted to discuss or publish trial results.